CLINICAL TRIAL: NCT01948973
Title: A Randomised, Controlled Crossover Study of Subsensory Sacral Nerve Stimulation for Irritable Bowel Syndrome
Brief Title: Subsensory Sacral Nerve Stimulation for Irritable Bowel Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 1-10-72-170-13, JLF; 1-10-72-170-13 (Other: VEK)
Record Dates: First submitted 2013-09-11; First posted 2013-09-24 (Estimated); Last update posted 2018-05-17 (Actual); Status verified 2018-05

CONDITIONS: Irritable Bowel Syndrome
Keywords: Irritable Bowel Syndrome; Sacral Nerve Stimulation; Symptoms; Quality of Life; Bowel habits
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- OFF, subsensory, suprasensory (Active Comparator): Here the stimulator is turned OFF for the first 2 weeks, then set subsensory (90% of sensory threshold) for the next 2 weeks and finally set suprasensory for the last 2 weeks.
  Interventions: Device: Subsensory; Device: OFF; Drug: Suprasensory
- Subsensory, OFF, suprasensory (Active Comparator): Here the stimulator is set subsensory (90% of sensory threshold), then turned OFF for the next 2 weeks and finally set suprasensory in the last 2 weeks.
  Interventions: Device: Subsensory; Device: OFF; Drug: Suprasensory

INTERVENTIONS:
Device: Subsensory — The stimulation is here set to 90% of the sensory threshold
  Other Names: Device: External pacemaker, model 3625, Medtronic Inc.
Device: OFF — The stimulation is here turned OFF
  Other Names: Device: External pacemaker, model 3625, Medtronic Inc.
Drug: Suprasensory — The stimulation is here set suprasensory
  Other Names: Device: External pacemaker, model 3625, Medtronic Inc.

SUMMARY:
Sacral nerve stimulation (SNS) has become a well-established treatment for patients with fecal incontinence since 1995. The mechanism of action of SNS is still not fully understood but recent studies have shown changes in both colonic motility and rectal sensibility. We have previously shown IBS patients to benefit from sacral nerves stimulation. With the present study, we aim to evaluate if subsensory sacral nerve stimulation is as effective as suprasensory sacral nerve stimulation.

DETAILED DESCRIPTION:
Twenty four patients with IBS-D or IBS-M according to the ROME III criteria, will be enrolled in the study.

Having meet inclusion criteria, the patients are randomised to receive either OFF-subsensory or subsensory-OFF stimulation in a 2+2-week period followed by 2 weeks of suprasensory stimulation. Hereby rendering a percutaneous nerve evaluation (PNE) test of a total of 6 weeks.

During the PNE test the effect of the stimulation is evaluated by specific IBS symptom and quality of life questionnaires (GSRS-IBS and IBS-IS) and bowel habit diaries.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged over 18
* Patients who are psychologically stable and suitable for intervention and able to provide informed consent.
* Patients who are diagnosed with IBS-D or IBS-M according to the Rome III criteria
* Minimum average of 40 points in the symptom quistionnaire evaluated at baseline

Exclusion Criteria:

* Overt bowel diseases including inflammatory bowel disease
* Pregnant or breast feeding
* Patients who are considered unable to follow the planned programme of the study, including mentally illness or physiological instability
* Patients who are on medication with known influence on gastrointestinal motility including those for thyroid disease, diabetes mellitus, celiac disease and neurological disease

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2013-09; Primary Completion 2018-03 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
The Gastrointestinal Symptom Rating Scale - Irritable Bowel Syndrome version questionnaire | Every week during the 6 weeks test period
  The GRSRS-IBS questionnaire is filled in every week during the test period allowing comparison between OFF, subsensory and suprasensory stimulation

SECONDARY OUTCOMES:
Irritable Bowel Syndrome - Impact Scale questionnaire | Every week during the 6 weeks test period
  The IBS-IS questionnaire is filled in every week during the test period allowing comparison of quality of life between OFF, subsensory and suprasensory stimulation

OTHER OUTCOMES:
Bowel habit diary | Every day during the 6 weeks test period
  The bowel habit diary is filled in every day during the test period allowing comparison between OFF, subsensory and suprasensory stimulation

CONTACTS AND LOCATIONS:
Overall Officials: Janne Fassov, PhD, Principal Investigator — Surgical Research Unit, Department of Surgery P, Aarhus University Hospital
Locations (1):
- Surgical Research Unit, Department of Surgery P, Aarhus University Hospital, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Fassov J, Hoyer KL, Lundby L, Laurberg S, Scott SM, Krogh K. Long-term efficacy and safety of sacral neuromodulation for diarrhoea-predominant and mixed irritable bowel syndrome. Tech Coloproctol. 2025 Jan 4;29(1):41. doi: 10.1007/s10151-024-03066-3. PMID 39754648